CLINICAL TRIAL: NCT03373786
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Pharmacodynamics, and Pharmacokinetics of RG-012 for Injection, Including Its Effect on Renal microRNA-21, in Subjects With Alport Syndrome
Brief Title: A Study of RG-012 in Subjects With Alport Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PDY16327; RG012-06 (Other: Regulus Therapeutics Inc.)
Record Dates: First submitted 2017-10-22; First posted 2017-12-14 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Alport Syndrome
Keywords: Kidney disease; Nephritis; Hereditary kidney disease; Hereditary nephritis
MeSH Terms: conditions — Nephritis, Hereditary; Kidney Diseases; Nephritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RG-012 Single Dose (Experimental): 1.5 mg/kg RG012 subcutaneous injection
  Interventions: Drug: RG012
- RG012 Every Other Week (Experimental): 1.5 mg/kg RG012 subcutaneous injections every other week
  Interventions: Drug: RG012

INTERVENTIONS:
Drug: RG012 — RG012 in 0.3% sodium chloride

SUMMARY:
This is a Phase 1, open-label, multi-center study of the safety, pharmacodynamics, and pharmacokinetics of RG-012 administered to subjects with Alport syndrome.

DETAILED DESCRIPTION:
This is a Phase 1, multi-center study of the safety, pharmacodynamics, and pharmacokinetics of RG-012 administered to subjects with Alport syndrome. During this open-label study, all eligible subjects will receive RG-012. The study consists of two parts (Part A and Part B). During Part A, half of the participants will receive a single dose of RG-012 and half will receive 4 doses of RG-012 (one dose every other week for 6 weeks). All subjects will undergo two renal biopsies, one before and one after receiving RG-012, to assess the effect of RG-012 on the kidney. After completing Part A, subjects will be able to enter Part B of the study. During Part B, all subjects will receive RG-012 every other week for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ages 18 to 65 years
2. Confirmed diagnosis of Alport syndrome
3. eGFR between 40 and 90 mL/min/1.73m2
4. Proteinuria of at least 300 mg protein/g creatinine
5. For subjects taking an ACE inhibitor or an ARB, the dosing regimen should be stable for at least 30 days prior to screening
6. Willing to comply with contraception requirements

Exclusion Criteria:

1. Causes of chronic kidney disease aside from Alport syndrome (such as diabetic nephropathy, hypertensive nephropathy, lupus nephritis, or IgA nephropathy)
2. End stage renal disease (ESRD) as evidenced by ongoing dialysis therapy or history of renal transportation
3. Any other condition that may pose a risk to the subject's safety and well-being
4. Female subjects who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse Events | 8 weeks
  Incidence and severity of adverse events
Effect of RG-012 on renal microRNA-21 (miR-21) | 8 weeks
  Change in miR-21 expression in renal tissue

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter - Cmax | 8 weeks
  Maximum observed plasma concentration
Pharmacokinetic (PK) parameter - Tmax | 8 weeks
  Time to maximum observed plasma concentration
Pharmacokinetic (PK) parameter - AUC | 8 weeks
  Area under the plasma concentration vs. time curve

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, M.D., Study Director — Sanofi
Locations (7):
- United States (7):
  - eStudySite, La Mesa, California
  - Academic Medical Research Institute, Los Angeles, California
  - Apex Research of Riverside, Riverside, California
  - Eminence Medical & Clinical Research, Tampa, Florida
  - Houston Nephrology Research, Cypress, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org